CLINICAL TRIAL: NCT06391866
Title: Assessing Neuroinflammation and Oxidative Stress After Cardiac Surgery: Unveiling Molecular Dynamics and Clinical Outcomes
Brief Title: Neuroinflammation/Oxidative Stress/Cardiac Surgery
Acronym: NEuOX-postSURg
Status: Recruiting | Type: Observational
Sponsor: Europainclinics z.ú. (Other)
Collaborators: East Slovak Institute for Cardiovascular Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: NeuOX-postSurg Trial
Record Dates: First submitted 2024-04-17; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Neuroinflammation
MeSH Terms: conditions — Neuroinflammatory Diseases | interventions — Extracorporeal Circulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental group 1: Patients scheduled for elective cardiac surgery, such as coronary artery bypass grafting (CABG) or valve replacement, involving extracorporeal circulation (ECC) with a duration less than 60 minutes.
  Interventions: Other: extracorporeal circulation
- Experimental group 2: Patients undergoing scheduled cardiac procedures, including coronary artery bypass grafting (CABG) or valve replacement, requiring extracorporeal circulation (ECC) for more than 60 minutes.
  Interventions: Other: extracorporeal circulation
- Control group:: Patients scheduled for cardiac surgical procedures such as coronary artery bypass grafting (CABG) without extracorporeal circulation, and for carotid endarterectomy in neurologically asymptomatic patients prior to the procedure.

INTERVENTIONS:
Other: extracorporeal circulation — extracorporeal circulation during cardiosurgical operation
  Groups: Experimental group 1; Experimental group 2

SUMMARY:
The prospective observational study delves into the complex relationship between neuroinflammation and oxidative stress in post-cardiac surgery complications, focusing on postoperative cognitive dysfunction.

DETAILED DESCRIPTION:
The prospective observational study meticulously examines the interplay between neuroinflammation and oxidative stress in the realm of post-cardiac surgery complications, specifically targeting postoperative cognitive dysfunction. Its primary objective is to comprehensively assess the sustained influence of these intricate processes on cognitive function and overall well-being, extending beyond the immediate aftermath of surgery. The research endeavors to probe deeply into the molecular mechanisms and clinical ramifications associated with neuroinflammation and oxidative stress, centering on their pivotal role in shaping the onset and trajectory of postoperative cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiosurgical operation
* Absence of previous neurological disease
* Signed informed consent document

Exclusion Criteria:

* Presence of neoplasms
* Neurological Disease
* Refusal to participate in the clinical trial

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patient undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number and type of early complications after surgery | 1 month
  Estimating of postoperative complications
Number and type of postoperative complications | 6 months
  Estimating of postoperative complications

SECONDARY OUTCOMES:
Estimating biochemical parameters | 1 hour
  Pro-inflammatory interleukins parameters (e.g. IL-8, IL-6, MIP-1a, MMP-2, MMP-9, SIRT 1, SIRT 2)
Estimating biochemical parameters | 6 hours
  Pro-inflammatory interleukins
Estimating biochemical parameters Third biochemical examination | 1 hour
  Antioxidative enzymes
Estimating biochemical parameters | 6 hours
  Antioxidative enzymes

CONTACTS AND LOCATIONS:
Locations (1):
- Europainclinics, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided
After completing data collection, the data will be made available to the ethical committees of interested institutions

REFERENCES:
- [Derived] Kocan L, Sudzina R, Kocanova H, Zavacka M, Pobehova J, Rybar D, Dudova M, Ferencik M, Vaskova J. Early Cognitive Outcomes After Carotid Endarterectomy in Asymptomatic Stenosis: A Pilot Study. Cureus. 2025 Nov 11;17(11):e96559. doi: 10.7759/cureus.96559. eCollection 2025 Nov. PMID 41393743